CLINICAL TRIAL: NCT02793128
Title: A Phase 3 Multicenter Trial Evaluating the Efficacy and Safety of UGN-101 on Ablation of Upper Urinary Tract Urothelial Carcinoma
Brief Title: The OLYMPUS Study - Optimized DeLivery of Mitomycin for Primary UTUC Study
Acronym: Olympus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC-UT-03-P
Record Dates: First submitted 2016-05-29; First posted 2016-06-08 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Carcinoma, Transitional Cell; Transitional Cell Carcinoma of Renal Pelvis
Keywords: TC-3; UTUC; Ureteral; Upper Tract; Carcinoma; Kidney; Renal; Gel; Local; Mitomycin C; Prolonged Release; Slow Release; Kidney Sparing; T1; T0; Low Grade; Transitional Cell Carcinoma of Renal Pelvis; TCC; UGN-101
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UGN-101 instillations (Experimental): The Mitomycin C (MMC) concentration of UGN-101 to be used in this trial will be 4 mg MMC per 1 mL of TC-3 gel, maximum dose is 15ml. 6 once weekly intravesical instillations for the ablation treatment.
  Interventions: Drug: UGN-101 instillations

INTERVENTIONS:
Drug: UGN-101 instillations — Treatment with UGN-101 once weekly for a total of 6 times; in a retrograde fashion. Patients who will demonstrate complete response (CR) will be treated with UGN-101 once monthly as a maintenance therapy for a total of 11 instillations or up to the first recurrence whichever comes first.
  Other Names: UGN-101

SUMMARY:
The study is investigating the ability of UroGen's UGN-101 to treat urothelial carcinoma tumors from the upper urinary tract.

DETAILED DESCRIPTION:
Trial TC-UT-03 is a prospective, open label, single-arm trial, designed to assess the efficacy, safety, and tolerability of treatment with UGN-101 instilled in the upper urinary system of patients with non-invasive low-grade (LG), Upper Tract Urothelial Carcinoma (UTUC).

Upon signing of informed consent, the patients will undergo a screening visit for eligibility evaluation. Eligible patients will be treated with UGN-101 once weekly for a total of 6 times; in a retrograde fashion. Patients who will demonstrate complete response (CR) will be treated with UGN-101 once monthly as a maintenance therapy for a total of 11 instillations or up to the first recurrence whichever comes first.

Five (5) weeks (± 1 w) following the last instillation, the Primary Disease Evaluation (PDE) Visit, during which safety and efficacy will be assessed, will take place. During this visit, the ablative effect of the UGN-101 will be assessed visually, by upper tract washed urine cytology, and if there are remaining tumors, by biopsy or brush biopsy if technically feasible.

Patient demonstrating CR at PDE will undergo monthly maintenance instillations of UGN-101 up to 11 months post PDE. Safety follow-up for these patients will be done until one month post last instillation or at the end of the follow-up period in FU visit 12, which is the earlier.

For patients who did not demonstrate Complete Response, to the extent that it is possible, all remaining tumors lesions will be biopsied. The patients shall undergo any additional surgical or other treatment the Principal Investigator (PI) decides deem necessary to remove remaining tumor.

An independent Data Monitoring Committee (DMC) was assigned to this trial. Accumulating safety, tolerability and efficacy data will be monitored periodically by the DMC according to a pre-specified process and frequency detailed in the DMC charter.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patient is at least 18 years of age.
2. Naive or recurrent patients with low grade (LG), non-invasive Upper Tract Urothelial Carcinoma (UTUC) in the pyelocalyceal system.
3. Patient has at least one (1) measurable papillary LG tumor, evaluated visually, ≤ 15 mm. The largest lesion should not exceed 15mm.
4. Biopsy taken from one or more tumors located above the ureteropelvic junction (UPJ) showing LG urothelial carcinoma. Diagnosed not more than 2 months prior to the screening.
5. Patient should have at least one remaining papillary LG tumor evaluated visually with a diameter of at least 5 mm.
6. Wash urine cytology sampled from the pyelocalyceal system documenting the absence of High Grade (HG) urothelial cancer, diagnosed not more than 2 months prior to the screening.
7. Patient with bilateral LG UTUC may be enrolled if at least one side meets the inclusion criteria for the trial and if the other kidney does not require further treatments (The other kidney can be treated prior to the beginning of the study).

Main Exclusion Criteria:

1. Patient received Bacille de Calmette et Guérin (BCG) treatment for Urothelial carcinoma (UC) during the 6 months prior to Visit 1.
2. The patient has untreated concurrent urothelial cancer in other locations other than the target area (unless treated during screening)
3. Carcinoma in situ (CIS) in the past in the urinary tract.
4. Patient has a history of invasive urothelial carcinoma in the urinary tract during the past 5 (Five) years.
5. Patient has a history of high grade papillary urothelial carcinoma in the urinary tract during the past 2 (Two) years.
6. Patient is actively being treated or intends to be treated with systemic chemotherapy during the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Lerner, M.D., Study Chair — Baylor College of Medicine
Locations (24):
- United States (22):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Loma Linda Cancer Center, Loma Linda, California
  - University of California, Los Angeles, California
  - Providence Medical Institute, Santa Monica, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Loyola University Medical Center, Department of Urology, Maywood, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - John Hopkins University, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic health system, Rochester, Minnesota
  - Urology Center Las Vegas, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center (Albert Einstein), The Bronx, New York
  - University of north carolina - chapel hill, Chapel Hill, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Thomas Jefferson University Hospitals, Philadelphia, Pennsylvania
  - MD Anderson, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Cancer Care Alliance (University of Washington), Seattle, Washington
- Israel (2):
  - Hasharon Hospital (Rabin Medical Center), Petah Tikva
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pierorazio PM, Kleinmann N, Shabsigh A, Hu B, Raman JD, Kaimakliotis H, Sankin A, Singla N, Meads A, Burger B, Raju S, Louie MJ, Chamie K, Weizer A, Schoenberg M. Long-Term Outcomes of Primary Chemoablation of Low-Grade Upper Tract Urothelial Carcinoma With UGN-101, a Mitomycin Reverse Thermal Gel. J Urol. 2025 Mar;213(3):313-322. doi: 10.1097/JU.0000000000004331. Epub 2024 Nov 19. PMID 39561384
- [Derived] Shabsigh A, Kleinmann N, Smith AB, Scherr D, Seltzer E, Schoenberg M, Lerner SP. Pharmacokinetics of UGN-101, a mitomycin-containing reverse thermal gel instilled via retrograde catheter for the treatment of low-grade upper tract urothelial carcinoma. Cancer Chemother Pharmacol. 2021 Jun;87(6):799-805. doi: 10.1007/s00280-021-04246-w. Epub 2021 Mar 7. PMID 33677615
- [Derived] Kokorovic A, Matin SF. UGN-101 (mitomycin gel): a novel treatment for low-grade upper tract urothelial carcinoma. Ther Adv Med Oncol. 2020 Jul 3;12:1758835920937950. doi: 10.1177/1758835920937950. eCollection 2020. PMID 32670424
- [Derived] Kleinmann N, Matin SF, Pierorazio PM, Gore JL, Shabsigh A, Hu B, Chamie K, Godoy G, Hubosky S, Rivera M, O'Donnell M, Quek M, Raman JD, Knoedler JJ, Scherr D, Stern J, Weight C, Weizer A, Woods M, Kaimakliotis H, Smith AB, Linehan J, Coleman J, Humphreys MR, Pak R, Lifshitz D, Verni M, Adibi M, Amin MB, Seltzer E, Klein I, Konorty M, Strauss-Ayali D, Hakim G, Schoenberg M, Lerner SP. Primary chemoablation of low-grade upper tract urothelial carcinoma using UGN-101, a mitomycin-containing reverse thermal gel (OLYMPUS): an open-label, single-arm, phase 3 trial. Lancet Oncol. 2020 Jun;21(6):776-785. doi: 10.1016/S1470-2045(20)30147-9. Epub 2020 Apr 29. PMID 32631491

RESULTS

PARTICIPANT FLOW:
Groups:
- UGN-101 Mitomycin for Pyelocalyceal Solution: This was a prospective, open-label, single-arm, pivotal phase study, designed to assess the efficacy, tolerability, and safety UGN-101 treatment administered to the Upper Urinary Tract (UUT).
  Upon signing of informed consent, the patients underwent a Screening Visit for eligibility evaluation.
  Eligible patients with confirmed low grade (LG) noninvasive Upper Tract Urothelial Carcinoma (UTUC) were treated with 6 once-weekly instillations of UGN-101. Tumor response was evaluated at the Primary Disease Evaluation (PDE) Visit, 5 weeks after the last treatment period instillation. Patients who demonstrated complete response (CR) could enter a maintenance period and receive up to 11 once-monthly instillations, per investigator modified treatment regimen.
Period: Overall Study
Arm/Group | UGN-101 Mitomycin for Pyelocalyceal Solution
Started | 71
Completed | 62
Not Completed | 9
Not completed — Death | 4
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Comorbid conditions and noncompliance | 1
Not completed — Patient elected nephroureterectomy | 1

BASELINE CHARACTERISTICS:
Groups:
- UGN-101 Mitomycin for Pyelocalyceal Solution: This was a prospective, open-label, single-arm, pivotal phase study, designed to assess the efficacy, tolerability, and safety UGN-101 treatment administered to the UUT. Upon signing of informed consent, the patients underwent a Screening Visit for eligibility evaluation.
  Eligible patients with confirmed LG noninvasive UTUC were treated with 6 once-weekly instillations of UGN-101. Tumor response was evaluated at the PDE Visit, 5 weeks after the last treatment period instillation. Patients who demonstrated CR could enter a maintenance period and receive up to 11 once-monthly instillations, per investigator modified treatment regimen.
Arm/Group | UGN-101 Mitomycin for Pyelocalyceal Solution
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 53
Age, Continuous [Median (Full Range); unit: years] | 71 [42 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 62
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 57
  Israel | 14

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint Was the Number of Patients Attaining Complete Response (CR) at the End of the Treatment Period (PDE Visit).
Description: The primary efficacy endpoint was the number of patients attaining complete response (CR) at the end of the treatment period (Primary Disease Evaluation (PDE) visit). The CR was defined dichotomously as "Success" if CR was confirmed at PDE visit (or relevant follow-up), and "Failure" otherwise.
Time Frame: An average of 11 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-101 Mitomycin for Pyelocalyceal Solution
Number analyzed (Participants) | 71
Participants | 42

2. Secondary Outcome: The Key Secondary Efficacy Endpoint Was Long-term Durability of Complete Response (CR): Number of Patients Who Maintained CR at 12 Month Post PDE Visit. This Endpoint Was Defined Only for Those Patients Who Achieved CR at the PDE Visit.
Description: Continuously: Duration of CR or time-to-recurrence since the Primary Disease Evaluation (PDE) Visit (i.e., time in days from the visit at which CR was determined until recurrence or censoring). This endpoint served as the main long-term durability endpoint. Dichotomously: "Success" if CR was still present at the 12 month post-PDE Visit (at Follow-Up Visit 4), and "Failure" otherwise. This endpoint served as a supportive long-term durability endpoint.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- UGN-101 Mitomycin for Pyelocalyceal Solution: Population was analyzed at 12 months post Primary Disease Evaluation (PDE) visit. 8 out of 41 patients had disease recurrence. The Kaplan-Meier estimate of 12 month duration of complete response (CR) rate was 82%.
  This was a prospective, open-label, single-arm, pivotal phase study, designed to assess the efficacy, tolerability, and safety UGN-101 treatment administered to the Upper Urinary Tract (UUT).
  Upon signing of informed consent, the patients underwent a Screening Visit for eligibility evaluation.
  Eligible patients with confirmed low grade (LG) noninvasive Upper Tract Urothelial Carcinoma (UTUC) were treated with 6 once-weekly instillations of UGN-101. Tumor response was evaluated at the PDE Visit, 5 weeks after the last treatment period instillation. Patients who demonstrated CR could enter a maintenance period and receive up to 11 once-monthly instillations, per investigator modified treatment regimen.
Arm/Group | UGN-101 Mitomycin for Pyelocalyceal Solution
Number analyzed (Participants) | 41
Participants | 23

3. Secondary Outcome: Durability of Complete Response (CR) for Each Follow-up Time Point.
Description: Durability of CR defined dichotomously as "Success" if CR was achieved at Primary Disease Evaluation (PDE) visit and remained at follow-up Visit 1, Visit 2 and Visit 3 (3, 6, 9 and 12 months post PDE visit), and "Failure" otherwise.
Time Frame: 3, 6, 9 and 12 months
Measure: Count of Participants; unit: Participants
Groups:
- UGN-101 Patients Evaluated 3 Months Post PDE: Patients reaching CR at PDE evaluated at 3 months post PDE
- UGN-101 Patients Evaluated at 6 Months Post PDE: Patients reaching CR at PDE evaluated at 6 months post PDE
- UGN-101 Patients Evaluated at 9 Months Post PDE: Patients reaching CR at PDE evaluated at 9 months post PDE
- UGN-101 Patients Evaluated at 12 Months Post PDE: Patients reaching CR at PDE evaluated at 12 months post PDE
Arm/Group | UGN-101 Patients Evaluated 3 Months Post PDE | UGN-101 Patients Evaluated at 6 Months Post PDE | UGN-101 Patients Evaluated at 9 Months Post PDE | UGN-101 Patients Evaluated at 12 Months Post PDE
Number analyzed (Participants) | 38 | 38 | 35 | 31
Participants | 35 | 33 | 28 | 23

4. Secondary Outcome: Clinical Benefit for Patients With Partial Response (PR) at the Primary Disease Evaluation (PDE) Visit. Clinical Benefit Endpoint Was Analyzed Using the Intent-to-Treat (ITT) Analysis Set, Including Patients Who Achieved Partial Response at PDE Visit.
Description: Clinical benefit for patients with partial response (PR) at the PDE visit. Clinical benefit endpoint was analyzed using the Intent-to-Treat (ITT) Analysis Set, including patients who achieved partial response at PDE Visit.Partial response at PDE visit will be defined dichotomously, similarly to the primary efficacy endpoint. For subjects with partial response at PDE visit, originally planned and actual treatments will be compared.
Time Frame: An average of 11 weeks
Measure: Count of Participants; unit: Participants
Groups:
- UGN-101 Mitomycin for Pyelocalyceal Solution: This was a prospective, open-label, single-arm, pivotal phase study, designed to assess the efficacy, tolerability, and safety UGN-101 treatment administered to the UUT.
  Upon signing of informed consent, the patients underwent a Screening Visit for eligibility evaluation.
  Eligible patients with confirmed LG noninvasive UTUC were treated with 6 once-weekly instillations of UGN-101. Tumor response was evaluated at the PDE Visit, 5 weeks after the last treatment period instillation. Patients who demonstrated CR could enter a maintenance period and receive up to11 once-monthly instillations, per investigator modified treatment regimen.
Arm/Group | UGN-101 Mitomycin for Pyelocalyceal Solution
Number analyzed (Participants) | 71
Participants | 8

5. Secondary Outcome: Pharmacokinetic: The PK Profiles of the First UGN-101 Instillation in the Blood Were to be Examined for the First 6 Patients.
Description: Cmax: maximum plasma concentration
  Analysis of individual plasma concentration versus time profiles showed that at 6 hours post instillation, the plasma concentrations of all 6 patients were below 2 ng/mL, with the plasma concentration of one patient dropping below the LOQ (i.e., < 0.100 ng/mL). The mean Cmax was 6.24 ng/mL (range: 2.43 to 12.80 ng/mL). The highest individual observed Cmax value of 12.80 ng/mL was 187-fold and 40 fold lower than the observed Cmax level following an intravenous bolus dose of 30 mg or 10 mg mitomycin (2.4 μg/mL and 0.52 μg/mL, respectively) and is 31 fold lower than the threshold value of 400 ng/mL for myelosuppression observed with mitomycin.
Time Frame: Blood samples were collected at 0 minutes (pre-dose) and 30 minutes, 1, 2, 3, 4, 5, and 6 hours following the first instillation of UGN-101
Population: PK Analysis Set: Consisted of patients who signed consent for PK and had sufficient PK data for the determination of PK parameters.
Measure: Mean (Inter-Quartile Range); unit: ng/mL
Groups:
- Pharmacokinetic Population: The PK profiles of the first UGN-101 instillation in the blood were to be examined for the first 6 patients.
Arm/Group | Pharmacokinetic Population
Number analyzed (Participants) | 6
ng/mL | 6.24 [2.43 to 12.80]

6. Other Pre Specified Outcome: Safety Adverse Event Outcomes: Safety Was Monitored Throughout the Study by Reviewing Adverse Events (AEs).
Description: Treatment-emergent AEs were most frequently reported from the Renal and urinary disorders system organ class (SOC), 59 (83.1%) patients, as expected, given the underlying indication of low grade (LG) Upper tract urothelial carcinoma (UTUC) in the study population, chemotherapeutic drug in a gel matrix instilled in the upper urinary tract (UUT), and the study procedure of treatment instillation via a ureteral catheter. The toxicity within the upper urinary tract was considered consistent with the disease under study and the mode of administration of UGN-101. Most events in the Renal and urinary disorders SOC were mild to moderate in severity and resolved. No new risks were identified and the overall safety profile was consistent with the known safety profile of endoscopic administration of intravesical mitomycin and of mitomycin. Overall, based on the safety and efficacy results to date, the benefit-risk profile of UGN-101 is favorable for the treatment of LG-UTUC.
Time Frame: Through study completion, an average of 15 months
Population: Safety: Consisted of all patients who enrolled in the study and received at least 1 instillation of UGN-101.
Measure: Count of Participants; unit: Participants
Groups:
- UGN-101 Mitomycin for Pyelocalyceal Solution: This was a prospective, open-label, single-arm, pivotal phase study, designed to assess the efficacy, tolerability, and safety UGN-101 treatment administered to the Upper Urinary Tract (UUT).
  Upon signing of informed consent, the patients underwent a Screening Visit for eligibility evaluation.
  Eligible patients with confirmed low grade (LG) noninvasive Upper Tract Urothelial Carcinoma (UTUC) were treated with 6 once-weekly instillations of UGN-101. Tumor response was evaluated at the PDE Visit, 5 weeks after the last treatment period instillation. Patients who demonstrated complete response (CR) could enter a maintenance period and receive up to11 once-monthly instillations, per investigator modified treatment regimen.
Arm/Group | UGN-101 Mitomycin for Pyelocalyceal Solution
Number analyzed (Participants) | 71
Participants
  Treatment-emergent Adverse Events (TEAEs) | 67
  TEAEs related to study drug | 52
  TEAEs related to study procedure | 55
  TEAEs related to study drug or preocedure | 61
  Serious Adverse Events (SAE) | 28
  SAEs related to study drug or procedure | 19

7. Secondary Outcome: Pharmacokinetic: The PK Profiles of the First UGN-101 Instillation in the Blood Were to be Examined for the First 6 Patients.
Description: Tmax: time to maximum plasma concentration
  Analysis of individual plasma concentration versus time profiles showed that at 6 hours post instillation, the plasma concentrations of all 6 patients were below 2 ng/mL, with the plasma concentration of one patient dropping below the LOQ (i.e., < 0.100 ng/mL).
  The mean Cmax was 6.24 ng/mL (range: 2.43 to 12.80 ng/mL), and the Tmax was 1.79 hours (range: 0.50 to 5.17 hours) after instillation. The highest individual observed Cmax value of 12.80 ng/mL was 187-fold and 40 fold lower than the observed Cmax level following an intravenous bolus dose of 30 mg or 10 mg mitomycin (2.4 μg/mL and 0.52 μg/mL, respectively) and is 31 fold lower than the threshold value of 400 ng/mL for myelosuppression observed with mitomycin.
Time Frame: Blood samples were collected at 0 minutes (pre-dose) and 30 minutes, 1, 2, 3, 4, 5, and 6 hours following the first instillation with UGN-101
Population: as for outcome 5
Measure: Mean (Inter-Quartile Range); unit: Hours
Arm/Group | Pharmacokinetic Population
Number analyzed (Participants) | 6
Hours | 1.79 [.5 to 5.17]

8. Secondary Outcome: Pharmacokinetic: The PK Profiles of the First UGN-101 Instillation in the Blood Were to be Examined for the First 6 Patients.
Description: Half-life (t½): terminal half-life
  The mean apparent t½ following instillation of mitomycin into the upper urinary tract (UUT) was 1.27 hours (76 minutes), which was longer than the true t½ of mitomycin following a 30 mg bolus injection (mean t½ value of approximately 17 minutes). The apparent t½ demonstrates that UGN-101 dissolved gradually, resulting in prolonged exposure of mitomycin following local instillation into the UUT.
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Number; unit: Hours
Arm/Group | Pharmacokinetic Population
Number analyzed (Participants) | 6
Hours | 1.27

ADVERSE EVENTS:
Time Frame: The study period for Adverse Events (AEs) collection was defined from the Informed Consent Form (ICF) signature and up to 30 days following the last administration of investigational product unless the AE was suspected to be related to the study treatment or was a Serious Adverse Event, in such case the AE should be reported regardless to the timelines of the reporting period. Through study completion, an average of 15 months.
Groups:
- UGN-101 Mitomycin for Pyelocalyceal Solution: This was a prospective, open-label, single-arm, pivotal phase study, designed to assess the efficacy, tolerability, and safety UGN-101 treatment administered to the Upper Urinary Tract (UUT).
  Upon signing of informed consent, the patients underwent a Screening Visit for eligibility evaluation.
  Eligible patients with confirmed Low Grade (LG) noninvasive Upper Tract Urothelial Carcinoma (UTUC) were treated with 6 once-weekly instillations of UGN-101. Tumor response was evaluated at the Primary Disease Evaluation (PDE) Visit, 5 weeks after the last treatment period instillation. Patients who demonstrated complete response (CR) could enter a maintenance period and receive up to11 once-monthly instillations, per investigator modified treatment regimen.
Arm/Group | UGN-101 Mitomycin for Pyelocalyceal Solution
All-Cause Mortality (participants affected / at risk) | 5/71
Serious Adverse Events (participants affected / at risk) | 28/71
Other Adverse Events (participants affected / at risk) | 67/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UGN-101 Mitomycin for Pyelocalyceal Solution (N=71)
Ureteric stenosis (Renal and urinary disorders) | 5 (5)
Hyrdornephrosis (Renal and urinary disorders) | 4 (4)
Flank Pain (Renal and urinary disorders) | 3 (3)
Urosepsis (Renal and urinary disorders) | 3 (3)
Heamaturia (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pulmonary oedema (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aortic dissection (Vascular disorders) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Subdural haematoma (Vascular disorders) | 1 (1)
Syncope (Vascular disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Gangrene (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1)
Transitional cell cancer of renal pelvis and ureter metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UGN-101 Mitomycin for Pyelocalyceal Solution (N=71)
Ureteric stenosis (Renal and urinary disorders) | 31 (31)
Urinary tract infection (Renal and urinary disorders) | 23 (23)
Haematuria (Renal and urinary disorders) | 23 (23)
Flank Pain (Renal and urinary disorders) | 22 (22)
Nausea (Gastrointestinal disorders) | 18 (18)
Dysuria (Renal and urinary disorders) | 16 (16)
Renal impairment (Renal and urinary disorders) | 14 (14)
Vomiting (Gastrointestinal disorders) | 14 (14)
Abdominal Pain (Gastrointestinal disorders) | 14 (14)
Hydronephrosis (Renal and urinary disorders) | 13 (13)
Fatigue (General disorders) | 11 (11)
Anemia (Blood and lymphatic system disorders) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Pollakiuria (Renal and urinary disorders) | 10 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9)
Pyrexia (General disorders) | 9 (9)
Chills (General disorders) | 8 (8)
Asthenia (General disorders) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7)
Hypertension (Vascular disorders) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Headache (Nervous system disorders) | 5 (5)
urinary tract inflammation (Renal and urinary disorders) | 5 (5)
Urinary tract obstruction (Renal and urinary disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Depression (Psychiatric disorders) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Renal Failure (Renal and urinary disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
urine abnormality (Renal and urinary disorders) | 4 (4)
Weight loss poor (Metabolism and nutrition disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2018-11-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02793128/ICF_001.pdf
  • Study Protocol (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02793128/Prot_003.pdf
  • Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT02793128/SAP_004.pdf